CLINICAL TRIAL: NCT03260790
Title: Immunogenicity of PPSV-23 After PCV-13 Vaccination in Adult Asthmatic Patients
Brief Title: Pneumococcal Vaccines in Patients With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Avni Joshi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-007731
Record Dates: First submitted 2017-07-31; First posted 2017-08-24 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Vaccine; Pneumococcal; Pneumonia
MeSH Terms: conditions — Asthma; Pneumonia | interventions — Heptavalent Pneumococcal Conjugate Vaccine; 23-valent pneumococcal capsular polysaccharide vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCV13 and PPSV23 (Experimental): Participants randomized to receive PPSV23 primed with PCV13. Participants will receive PCV13 8 weeks prior to receiving PPSV23
  Interventions: Biological: PCV13; Biological: PPSV23
- PPSV23 (Active Comparator): Participants randomized to receive PPSV23 alone
  Interventions: Biological: PPSV23

INTERVENTIONS:
Biological: PCV13 — Single 0.5 ml dose of PCV13 administered via intramuscular injection
  Other Names: Prevnar
  Arms: PCV13 and PPSV23
Biological: PPSV23 — Single 0.5 ml dose of PPSV23 administered via intramuscularly or subcutaneously
  Other Names: Pneumovax

SUMMARY:
Investigators are assessing if patients with asthma respond better to the Pneumovax vaccine if they are given Prevnar initially.

DETAILED DESCRIPTION:
Patients will be randomized into either PCV13 and PPSV23 (Experimental) or PPSV23 alone (Active comparator). At the Week 0 time point, the patients will receive either PCV13 (Experimental) or PPSV23 (Active comparator) and undergo a blood draw of 5ml for assessment of pre-vacation serotype titers. The Active Comparator group will undergo a 5ml draw of blood for assessment of titers at week 8, 16, and 24 following vaccination. The Experimental group will undergo vaccination with PPSV23 at week 8 with 5 ml blood draw for pneumococcal serotype titers as well as a blood draw at week 16 and week 24.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of asthma

Exclusion Criteria:

* Research exemption requested
* History of PCV-13 vaccination
* History of cochlear implant
* Cerebrospinal Fluid (CSF) leak
* Congestive Heart Failure (CHF)
* Diabetes Mellitus (DM)
* Chronic Kidney Disease (CKD)
* Human Immunodeficiency Virus (HIV)
* Common Variable Immune Deficiency (CVID)
* Patients who have received the PPSV23 vaccine in the last 5 years
* Women who are pregnant will also be excluded from the study by performing 2 point of care urine pregnancy tests ( prior to vaccinations)

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avni Y Joshi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- PCV13 and PPSV23: Participants received PPSV23 primed with PCV13. Participants received PCV13 8 weeks prior to receiving PPSV23
  PCV13: Single 0.5 ml dose of PCV13 administered via intramuscular injection
  PPSV23: Single 0.5 ml dose of PPSV23 administered 8 weeks after receiving PCV13 via intramuscularly or subcutaneously
- PPSV23: Participants received PPSV23 alone
  PPSV23: Single 0.5 ml dose of PPSV23 administered via intramuscularly or subcutaneously
Period: Overall Study
Arm/Group | PCV13 and PPSV23 | PPSV23
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCV13 and PPSV23 | PPSV23 | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Total Anti-pneumococcal IgG Levels at Baseline, Week 0, Week 8 and Week 16
Description: 5 ml blood draw for assessment of pneumococcal specific titer IgG. Measured as mcg/dL.
Time Frame: Baseline, week 0, week 8, week 16
Population: Baseline = For arm PPSV23 baseline is 8 weeks prior to receiving PPSV-23. For arm PCV13 and PPSV23 baseline is day of receiving PCV-13. Week 0 = day of receiving PPSV-23 for both arms. Week 8 = eight weeks after receiving PPSV-23 for both arms. Week 16 = sixteen weeks after receiving PPSV-23 for both arms.
Measure: Median (Inter-Quartile Range); unit: mcg/dL
Arm/Group | PCV13 and PPSV23 | PPSV23
Number analyzed (Participants) | 8 | 9
mcg/dL
  baseline | 109.8 [74.3 to 141.8] | 53.9 [34.8 to 185.3]
  week 0 | 142.3 [111.7 to 194.6] | 53.9 [34.8 to 185.3]
  week 8 | 211.7 [184.6 to 271.0] | 243.3 [173.4 to 271.0]
  week 16 | 212.0 [171.1 to 257.7] | 224.8 [196.6 to 271.0]

2. Primary Outcome: Sum of Anti-pneumococcal IgG to All Serotypes at Baseline, Week 0, Week 8 and Week 16
Description: 5 ml blood draw for assessment of IgG specific Antibody titers to all 23 serotypes. Measured as mcg/mL.
Time Frame: Baseline, week 0, week 8, week 16
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mcg/mL.
Arm/Group | PCV13 and PPSV23 | PPSV23
Number analyzed (Participants) | 8 | 9
mcg/mL.
  baseline | 228.0 [174.2 to 362.3] | 206.8 [130.1 to 323.8]
  week 0 | 506.3 [349.6 to 670.9] | 206.8 [130.1 to 323.8]
  week 8 | 502.9 [369.9 to 790.5] | 449.4 [338.7 to 583.4]
  week 16 | 534.8 [325.4 to 688.4] | 485.7 [321.2 to 588.6]

3. Primary Outcome: Sum of Anti-pneumococcal IgG to Serotypes Common to PCV13 and PPSV23 at Baseline, Week 0, Week 8, Week 16
Description: 5 ml blood draw for assessment of IgG specific Antibody titers for serotypes common PCV13 & PPSV23. Measured as mcg/mL.
Time Frame: Baseline, week 0, week 8, week 16
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | PCV13 and PPSV23 | PPSV23
Number analyzed (Participants) | 8 | 9
mcg/mL
  baseline | 142.4 [110.7 to 246.8] | 107.4 [92.9 to 161.8]
  week 0 | 418.9 [303.2 to 525.1] | 107.4 [92.9 to 161.8]
  week 8 | 362.8 [258.9 to 498.6] | 229.4 [162.6 to 302.2]
  week 16 | 343.7 [221.5 to 447.1] | 230.5 [149.5 to 302.1]

4. Primary Outcome: Sum of Anti-pneumococcal IgG to Serotypes Unique to PPSV23 at Baseline, Week 0, Week 8 and Week 16.
Description: 5 ml blood draw for assessment of IgG specific Antibody titers for serotypes unique to PPSV23. Measured as mcg/mL.
Time Frame: Baseline, week 0, week 8, week 16
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | PCV13 and PPSV23 | PPSV23
Number analyzed (Participants) | 8 | 9
mcg/mL
  baseline | 89.2 [64.1 to 120.9] | 74.7 [41.0 to 160.2]
  week 0 | 82.4 [56.2 to 152.4] | 74.7 [41.0 to 160.2]
  week 8 | 174.2 [92.3 to 283.4] | 220.0 [164.7 to 246.8]
  week 16 | 179.1 [96.9 to 277.0] | 184.1 [171.0 to 255.2]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 16 weeks.
Groups:
- PCV13 and PPSV23: Participants received PPSV23 primed with PCV13
  PCV13: Single 0.5 ml dose of PCV13 administered via intramuscular injection
  PPSV23: Single 0.5 ml dose of PPSV23 administered 8 weeks after receiving PCV13 via intramuscularly or subcutaneously
Arm/Group | PCV13 and PPSV23 | PPSV23
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT03260790/Prot_SAP_000.pdf